CLINICAL TRIAL: NCT00556101
Title: Whole Body Magnetic Resonance Angiography: Questionnaire Examination of Patient Acceptance.
Brief Title: Patient Acceptance of Whole Body Magnetic Resonance Angiography
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital at Herlev (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Other Study IDs: WB-angio herlev 4
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Atherosclerosis; Intermittent Claudication; MRI
Keywords: Magnetic resonance; whole body; angiography; questionnaire
MeSH Terms: conditions — Atherosclerosis; Intermittent Claudication

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Whole body magnetic resonance angiography

SUMMARY:
Investigation of how the patients experience whole body MRA. After the WB-MRA the patients will fill in a questionnaire, that contains questions about the WB-MRA procedure and how the patient felt during the examination.

We expect that the patients will report a high degree of satisfaction with the WB-MRA procedure, with little discomfort.

DETAILED DESCRIPTION:
WB-MRA is performed in patients referred for conventional x-ray based angiography. The WB-MRA is performed first in all patients.

After both examinations are completed the patients will be asked to fill in a questionnaire containing questions about their experience of the 2 procedures.

We will then compare the results for the procedures.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic lower extremity ischemia (claudication, ischemic wounds)
* Referred to digital subtraction angiography (DSA)

Exclusion Criteria:

* Renal insufficiency (GFR < 30 ml/min)
* Contra-indications for MRI-examination (claustrophobia, metal-implants, pacemaker)
* Dementia
* Pregnancy/lactation
* Allergy to gadolinium based MRI contrast agents
* Acute disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pheripheral arterial disease
Sampling Method: Non-Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2007-11; Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Patient acceptance of Whole body MRA

CONTACTS AND LOCATIONS:
Overall Officials: Henrik S Thomsen, Prof. MD., Study Chair — University Hospital at Herlev Copenhagen Denmark
Locations (1):
- Department of Radiology, Herlev University Hospital, Herlev Copenhagen, Herlev, Denmark